CLINICAL TRIAL: NCT03183713
Title: The Confounding Burden of Psychological Impairments in Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-02144
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cervical Spine Disease; Psychological Impairment
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparison Group (Active Comparator): Patients with a zero risk score will serve as a comparison group (N=20).
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Sham Treatment (Active Comparator): All patients at risk will be stratified by risk rating and randomly assigned to 2 groups; sham treatment (N=20) or CBT (N=20).
  Interventions: Behavioral: Sham Therapy
- CBT (Active Comparator): All patients at risk will be stratified by risk rating and randomly assigned to 2 groups; sham treatment (N=20) or CBT (N=20).
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Psychologically symptomatic patients will then be randomized to 4-8 weeks of placebo phone calls (Group PS-PL-Sx) or 4-8 weeks of cognitive behavior therapy treatment (PS-CBT-Sx) based on a 1:1 randomization ratio. Subjects randomized to receive CBT before surgery will proceed to 6 sessions given within 4-8 weeks by a licensed psychologist specializing in pain. CBT sessions will be 30 minutes in length, and focus on empirically supported behavior management, problem solving, cognitive restructuring, and relaxation training. The first session will be performed in person, and the subsequent 5 sessions will be performed over the phone.
  Arms: CBT; Comparison Group
Behavioral: Sham Therapy — Study nurse will conduct six sessions (30 minutes/ session) over a 4-8 week time period. The first session will be performed in person, and the subsequent 5 sessions will be performed over the phone. Sham sessions will entail how to prepare for surgery and expectations for recovery, and will go over content that the treatment and control groups will receive in handout form.
  Arms: Sham Treatment

SUMMARY:
This is a single-center prospective randomized investigation of patients undergoing surgical arthrodesis for single or multi-level cervical disease, resulting in cervical radiculopathy. Patients indicated for surgery for cervical degenerative disease (CDD) will be screened for yellow flags using validated tools to assess pain. Cognitive-behavioral therapy (CBT) will be used to modify yellow flags in spine patients. All patients at risk will be stratified by risk rating and randomly assigned to 2 groups; sham treatment (N=20) or CBT (N=20). The goal of this study is to unmask the relationship between psychological distress and clinical outcomes in patients undergoing surgical treatment for cervical degenerative disease resulting in combinations of neck pain and radiculopathy, and to determine the effectiveness of a brief psychological intervention on subset of patients who screen positive for psychological distress prior to their surgeries.

ELIGIBILITY:
Inclusion Criteria:

Patients at Risk:

* Diagnosed of primary symptomatic cervical degenerative disc disease confirmed with appropriate imaging studies.
* Etiologies will be limited to cervical disc herniation, spinal stenosis, low-grade (I and II) spondylolisthesis, spondylosis and degenerative disc disease.
* Will be undergoing elective cervical spine surgery, not to exceed 5 levels.
* Presence of both axial (neck pain) and appendicular (arm pain/dysesthesia/weakness) symptoms, regardless of proportion
* Subject must be able to be contacted by telephone during study participation
* NDI > 20%
* Read and comprehend English

Inclusion Criteria for patients with zero risk:

* Diagnosed of primary symptomatic cervical degenerative disc disease confirmed with appropriate imaging studies.
* Etiologies will be limited to cervical disc herniation, spinal stenosis, low-grade (I and II) spondylolisthesis, spondylosis and degenerative disc disease.
* Will be undergoing elective cervical spine surgery, not to exceed 5 levels.
* Presence of both axial (neck pain) and appendicular (arm pain/dysesthesia/weakness) symptoms, regardless of proportion
* Subject must be able to be contacted by telephone during study participation
* NDI > 20%
* Read and comprehend English

Exclusion Criteria:

Exclusion Criteria for patients at risk:

* Contraindicated to surgical treatment of the cervical spine.
* Prior cervical fusion
* Evidence of severe cervical spinal deformity based on Ames classification: C2-C7 SVA > 8cm, Horizontal Gaze < -10 or > 25, T1S-CL > 20, myelopathy (JOA score <10) or severe adult spinal deformity based on SRS-Schwab classification (PI-LL > 20, PT >30, SVA > 90 mm)
* Undergoing simultaneous treatment for thoracolumbar spine related diagnoses at the time of enrollment History of any spinal surgery within the last 6 months
* Patients with neck pain attributable to trauma, idiopathic deformity, neoplasm, osteoporosis, or other medical condition.
* Unlikely to comply with the follow-up evaluation schedule
* Subject has recent history of chemical substance dependency that may impact the outcome or study participation

Exclusion Criteria for patients with zero risk:

* Contraindicated to surgical treatment of the cervical spine.
* Prior cervical fusion
* Evidence of severe cervical spinal deformity based on Ames classification: C2-C7 SVA > 8cm, Horizontal Gaze < -10 or > 25, T1S-CL > 20, myelopathy (JOA score <10) or severe adult spinal deformity based on SRS-Schwab classification (PI-LL > 20, PT >30, SVA > 90 mm)
* Undergoing simultaneous treatment for thoracolumbar spine related diagnoses at the time of enrollment History of any spinal surgery within the last 6 months
* Patients with neck pain attributable to trauma, idiopathic deformity, neoplasm, osteoporosis, or other medical condition.
* Unlikely to comply with the follow-up evaluation schedule
* Subject has recent history of chemical substance dependency that may impact the outcome or study participation
* Subject has a significant psychosocial disturbance or psychiatric history that may impact the outcome or study participation including a DRAM score over 33
* Active infection
* Systemic infection (AIDS, HIV, or active hepatitis)
* Active litigation
* Presence of inflammatory spinal disease (e.g. chronic autoimmune conditions, ankylosing spondylitis, DISH, Rheumatoid Arthritis)
* Concurrent Spinal or pelvic fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Distress and Risk Assessment Method (DRAM) | 2 Years
  The DRAM assesses and profiles patients: those showing no psychological distress, those at risk of developing major psychological overlay, and those that are distressed.
Pain Catastrophizing Scale (PCS) | 2 Years
  The pain catastrophizing scale quantifies an individual's pain experience, their tendency to magnify the threat value of pain, and their ability to prevent pain-related thoughts surrounding a painful event.
Outcome Expectation question (OEQ) | 2 Years
  The OEQ will be a single item question: "I strongly believe that I will recover quickly from my surgery. Responses are score on a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Outcome expectations have been shown to be one of the strongest psychological predictors affecting recovery from musculoskeletal injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Passias, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States